CLINICAL TRIAL: NCT06668051
Title: Determination of Functional Exercise Capacity, Peripheral Muscle Strength, Respiratory Muscle Endurance and Parameters Affecting Quality of Life in Idiopathic Pulmonary Fibrosis
Brief Title: Determination of Functional Exercise Capacity, Respiratory Muscle Endurance in Idiopathic Pulmonary Fibrosis
Status: Not yet recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Bilge Gore, physiotherapist, Hacettepe University
Other Study IDs: GO 23/14
Record Dates: First submitted 2024-09-16; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Idiopathic Pulmonary Fibrosis; Healthy
Keywords: Quality of life; Muscle strength; Respiratory function tests; Pulmonary fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- IPF: Inclusion Criteria: Being over 18 years old -having a clinical, radiological and/or pathological diagnosis of IPF -volunteering to participate in the study -not having had a respiratory tract infection in the last month -not having an accompanying airway disease such as COPD -being in the stable phase of the disease Exclusion Criteria: Patients who have had an IPF attack within the last three months and/or are in the acute exacerbation of the disease; who use a walking aid; who have unstable angina or class III-IV heart failure according to the New York Heart Association congestive heart failure classification; who have orthopedic, neuromuscular, neurological and cardiac diseases that may affect walking and balance; who have serious comorbid conditions such as cancer or neoplasm; who have a history of sarcoidosis, tuberculosis, emphysema and/or lung surgery; who have communication problems, mental and cognitive problems, and who cannot adapt to the applied assessment methods will be
- HEALTHY GROUP: Being over 18 years old -having a clinical, radiological and/or pathological volunteering to participate in the study -not having had a respiratory tract infection in the last month -not having an accompanying airway disease such as COPD

SUMMARY:
There are not enough studies in the literature comparing functional capacity, respiratory functions and muscle strength of IPF patients with healthy individuals. This study aims to compare functional capacity, respiratory functions and muscle strength of IPF patients with healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* having a clinical, radiological and/or pathological diagnosis of IPF
* volunteering to participate in the study
* not having had a respiratory tract infection in the last month
* not having an accompanying airway disease such as COPD
* being in the stable phase of the disease

Exclusion Criteria:

* Patients who have had an IPF attack within the last three months and/or are in the acute exacerbation of the disease; who use a walking aid; who have unstable angina or class III-IV heart failure according to the New York Heart Association congestive heart failure classification; who have orthopedic, neuromuscular, neurological and cardiac diseases that may affect walking and balance; who have serious comorbid conditions such as cancer or neoplasm; who have a history of sarcoidosis, tuberculosis, emphysema and/or lung surgery; who have communication problems, mental and cognitive problems, and who cannot adapt to the applied assessment methods will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 12 patients with IPF will be included in the patient group. Twelve healthy individuals, similar in age and gender to the patient group, will be included in the study as a control group.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2025-01-22 (Estimated); Study Completion 2025-02-22 (Estimated)

PRIMARY OUTCOMES:
6 Minute Walk Test (6MWT) | 1 month
  6 MWT is a submaximal test that evaluates the functional exercise capacity of individuals. Individuals will walk along a 30-meter corridor at their maximum speed. Individuals will be asked to walk as much distance as possible within the given time without running or jumping.The time will be started as soon as individuals start walking. Before and after the test, O2 saturation with pulse oximeter, heart rate, dyspnea and fatigue severity with Borg scale will be evaluated between 0 and 10 points (0; no symptoms, 10; most severe symptoms). Individuals will be asked to stop the test if they do not feel well during the test. When the time is up, participants will be asked to leave the sign given for marking purposes on the ground and the walking distance will be evaluated with the sign.
6 Minute Pegboard and Ring Test | 1 month
  This test will be used to measure upper extremity function. The test will be performed using a Pegboard with two upper and two lower pegs placed at the patients shoulder level and above shoulder level (20 cm). Ten rings will be placed on each lower peg. During the test, patients move each of the rings on the lower pegs to the upper pegs using both hands simultaneously, and then move the rings back from the upper pegs to the lower pegs. The goal is to move as many rings as possible for six minutes. The score will be reported as the number of rings moved simultaneously. Patients will be allowed to stop and rest during the test if they experience severe shortness of breath, fatigue, or other discomfort, and to resume moving the rings as soon as possible. Scores will be measured for heart rate, blood pressure, perception of dyspnea, and upper extremity fatigue before and immediately after each test.
30-second sit to stand test | 1 month
  This test reflects the strength of the lower extremities. The individual sits in the middle of a chair with no armrests and a sitting height of 43 cm, with his back straight and straight, his arms crossed in front, and his feet touching the floor. With the start command, he stands up and sits down completely. The individual who learns the test with a stopwatch is asked to sit down and stand up for 30 seconds and the score obtained is recorded as the number of repetitions in the evaluation form.
Forced Vital Capasity | 1 month
  Forced vital capacity (FVC) is the volume of air that is exhaled quickly and forcefully following a deep inspiration. It is a pulmonary function test parameter and performed using spirometry. The best value obtained from three technically acceptable measurements is expressed as a percentage of the expected value calculated from age, gender and height.
Respiratory Muscle Strength Assessment | 1 month
  Respiratory muscle strength will be determined by measuring the maximal inspiratory pressure (MIP) created in the mouth using a mouth pressure device and the maximum expiratory pressure (MEP) with personal antibacterial and antiviral disposable filters. During the MIP measurement, the patient is asked to make a maximum expiration, and the patient's nose is closed with a clip and then the patient's nose is closed with a clip and then the patient is asked to make a maximum inspiration for 1-3 seconds. During the MEP measurement, the patient is asked to make a maximum inspiration, and the patient's nose is closed with a clip and then the patient's nose is closed with a clip and then the patient's nose is closed with a clip and then the tests are repeated until no further improvement is observed and there is no difference of more than 5% between the 2 best values.
Respiratory Muscle Endurance Test | 1 month
  It is applied at 60% of maximal inspiratory pressure. After the device is placed in the mouth, the nose is closed with a clamp. The patient is asked to breathe in and out through the mouth for 10 minutes. Before starting the test, patients are informed that if they feel too much shortness of breath during the test, they can remove the device and the test will end in this way. Before and after the test, the SpO2 value is measured with a portable pulse oximeter attached to the finger; dyspnea perception is measured and recorded with the Modified Borg Scale.
Hand Grip Strength | 1 month
  A Jamar Hydraulic Hand Dynamometer (Jamar Hydraulic Hand Dynamometer, Cedarburg, England) will be used to measure hand grip strength. The Jamar hand dynamometer is considered the most reliable tool for measuring grip strength. Individuals are asked to sit with the shoulder adducted, the elbow flexed at 90°, the forearm in the middle position, and the wrist in a neutral position. Participants are asked to hold the handle and squeeze with the maximum force they can. The measurement begins with the dominant hand. Three consecutive measurements are taken for the dominant and non-dominant hands, with a 1-minute interval between measurements. The highest value of the three measurements is recorded.
Quadriceps Strength | 1 month
  Measurements will be made with a portable digital muscle strength tester (01165 manual muscle tester, Lafayette Instrument Co. Lafayette, USA) to evaluate knee extensor muscle strength. It will be applied while individuals are in a sitting position on the edge of the bed with their knees bent to 90° and the space between the back of the knee and the bed filled with a towel. Individuals are asked to cross their hands on their chest and sit with their bodies upright. When the test begins, the knee is bent and the knee is straightened. The researcher measures the knee extensor muscle strength by applying force slightly above the ankle and trying to push downward in order to overcome the straight knee force. The test is repeated three times to measure the right and left knee extensor muscle strength and the highest value obtained is recorded in kilograms (kg) and Newtons (N).
Respiratory Function Testing | 1 month
  It is performed using a spirometer. The best value obtained from three technically acceptable measurements is expressed as a percentage of the expected value calculated from age, gender and height. The patient must be in an upright sitting position during the test.
Forced expiratory volume in 1 second | 1 month
  forced expiratory volume in 1 second (FEV1) is the volume of air exhaled in the first second from the beginning of the forced vital capacity maneuver. In general, it provides information about the restriction in the large airways. It is a pulmonary function test parameter and performed using spirometry. The best value obtained from three technically acceptable measurements is expressed as a percentage of the expected value calculated from age, gender and height.
Forced expiratory flow between 25 and 75% of vital capacity (FEF 25-75) | 1 month
  Forced expiratory flow between 25 and 75% of vital capacity (FEF 25-75) is the average flow rate at 50% of the forced vital capacity maneuver. It provides information about the obstruction in medium and small bronchi. It is a pulmonary function test parameter and performed using spirometry. The best value obtained from three technically acceptable measurements is expressed as a percentage of the expected value calculated from age, gender and height.
Peak expiratory flow | 1 month
  Peak expiratory flow (PEF) is measured with a maximum inspiration followed by a maximum exhalation maneuver. It provides information about obstruction in the large airways. It is a pulmonary function test parameter and performed using spirometry. The best value obtained from three technically acceptable measurements is expressed as a percentage of the expected value calculated from age, gender and height.
FEV1/FVC | 1 month
  A low FEV1/FVC ratio (<80%) is used as a primary obstruction parameter. It is a pulmonary function test parameter and performed using spirometry. The best value obtained from three technically acceptable measurements is expressed as a percentage of the expected value calculated from age, gender and height.

SECONDARY OUTCOMES:
TAMPA KINESOPHOBIA SCALE | 1 month
  TAMPA KINESOPHOBIA SCALE is a 17-question scale developed to measure fear of movement/re-injury (150). The scale includes parameters of injury, re-injury and avoidance-fear in physical activities related to daily life and work. It is a Likert-type 4-point scale (1=strongly disagree, 2=disagree, 3=agree, 4=strongly agree). In this questionnaire, where a maximum score of 68 and a minimum score of 17 are obtained; a score greater than 37 is classified as high-degree kinesiophobia, and a score equal to or lower is classified as low-degree kinesiophobia.
LEICESTER COUGH QUESTIONNAIRE | 1 month
  The Leicester cough questionnaire is a short, easy-to-apply, valid questionnaire developed to investigate the effect of chronic cough on quality of life. It includes 3 areas and 19 topics: physical, psychological and social. In this questionnaire, patients answer the questions themselves; they select the topics they identify as problems and rank them according to the importance attributed to them. The topics are divided into areas using clinical logic. A seven-point Likert scale is used for evaluation.The score for each area is calculated by dividing the patient's total score for each question by the number of questions. The score for each area ranges from 1 to 7. The total score is the sum of the 3 areas (physical, psychological and social) The total score range is 3 to 7. A higher score indicates a better health status. .
St. George's Respiratory Questionnaire (SQRQ) | 1 month
  St. George's Respiratory Questionnaire (SQRQ): The effects of the disease on quality of life are examined in 3 sections: symptoms, activity and impact. SGRQ consists of 76 questions. It has a scale of 0 to 100 points. Zero indicates good health status, 100 indicates the worst disease status
Bouchard Three-Day Physical Activity Record | 1 month
  Bouchard Three-Day Physical Activity Record: Bouchard's physical activity diary is an example of a widely used activity record in which participants report their activities every 15 minutes. Activities are rated from 1 to 9 (1 = sedentary, 9 = vigorous/vigorous activity) to obtain a total energy expenditure score. The resulting numbers are added together and multiplied by the MET values to calculate the estimated daily energy expenditure (kcal/kg1).

IPD SHARING:
Plan to Share IPD: Undecided